CLINICAL TRIAL: NCT02025426
Title: Impact of Vasopressor Administration on Maternal and Neonatal Outcomes in Women With Pre-eclampsia
Brief Title: Phenylephrine Versus Ephedrine in Pre-eclampsia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant challenges recruiting a difficult patient population with most surgeries occurring out of hours
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00032812
Record Dates: First submitted 2013-12-26; First posted 2014-01-01 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Pre-eclampsia
Keywords: Cesarean delivery; Spinal Anesthesia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Phenylephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine (Active Comparator): Phenylephrine for maintaining blood pressure within 10 % of baseline
  Interventions: Drug: Phenylephrine
- Ephedrine (Active Comparator): Ephedrine for maintaining blood pressure within 10 % of baseline
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Phenylephrine
  Arms: Phenylephrine
Drug: Ephedrine
  Arms: Ephedrine

SUMMARY:
Phenylephrine administration is associated with reductions in CO and SctO2 compared with ephedrine when used for blood pressure management in women with pre-eclampsia undergoing cesarean delivery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age ≥18 yrs
* Pre-eclampsia (mild, or severe)
* Non-laboring women
* CD under spinal anesthesia

Exclusion Criteria:

* Height < 5'0"
* Allergy to phenylephrine or ephedrine, or any other standardized medication
* Severe Cardiac disease in pregnancy with marked functional limitations (NYHA Class III and IV)
* Patients on Monoamine Oxidase Inhibitors or Tricyclic Antidepressants
* History of recent amphetamine or cocaine use.
* Subject enrollment in another study involving a study medication within 30 days of CD
* Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenylephrine: Phenylephrine for maintaining blood pressure within 10 % of baseline
  Phenylephrine
- Ephedrine: Ephedrine for maintaining blood pressure within 10 % of baseline
  Ephedrine
Period: Overall Study
Arm/Group | Phenylephrine | Ephedrine
Started | 9 | 4
Completed | 9 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Ephedrine | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.89 (8.72) | 39.25 (10.14) | 32.77 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6 | 2 | 8
  Caucasian | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 4 | 13
Weight [Mean (Standard Deviation); unit: kg] | 107.76 (29.62) | 117.35 (27.26) | 110.71 (28.14)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 40.53 (11.58) | 44.55 (12.85) | 41.77 (11.59)
Height [Mean (Standard Deviation); unit: cm] | 163.22 (4.94) | 163.47 (6.47) | 163.30 (5.17)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 32.67 (4.42) | 35.25 (3.59) | 33.46 (4.22)
Gravida [Mean (Standard Deviation); unit: pregnancies] — The total number of confirmed pregnancies that a woman has had, regardless of the outcome.
  pregnancies | 3.00 (1.85) | 3.25 (1.26) | 3.08 (1.62)
Para [Mean (Standard Deviation); unit: births] — The number of births that a woman has had after 20 weeks gestation.
  births | 1.25 (1.04) | 1.50 (1.29) | 1.33 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Tissue Oxygen Saturation
Time Frame: Intraoperative from spinal placement till 10 min after delivery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
mmHg | 30.08 (29.32) | 19.10 (7.23)
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p = 0.547, Kruskal-Wallis

2. Secondary Outcome: Cardiac Output
Time Frame: Intraoperative from spinal placement till 10 min after delivery
Population: Data for cardiac output from Physioflow worksheets was not available for two participants in the Phenylephrine group and all four participants in the Ephedrine group.
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 7 | 0
mL/minute | 8.19 (4.76) |

3. Other Pre Specified Outcome: Neonatal Umbilical Cord Gases, pCO2
Description: Partial pressure of carbon dioxide (pCO2) is the measure of carbon dioxide within arterial blood flowing through the umbilical cord.
Time Frame: Within 5 minutes after delivery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
mmHg | 56.71 (11.80) | 55.93 (12.97)
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p = 0.925, Kruskal-Wallis

4. Other Pre Specified Outcome: Neonatal Umbilical Cord Gases, pH
Description: Used to assess acid-base balance. pH ranges from 0 to 14 and a pH of 7.40 is considered standard (normal) conditions.
Time Frame: Within 5 minutes after delivery
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
unitless | 7.24 (0.07) | 7.19 (0.15)
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p = 0.498, Kruskal-Wallis

5. Other Pre Specified Outcome: Neonatal Umbilical Cord Gases, BE
Description: The amount of strong acid (in mmol/L) that needs to be added in vitro to 1 liter of fully oxygenated blood in order to return the sample to standard (normal) conditions (pH 7.40, pCO2 40 mmHg and temperature 37 °C.)
Time Frame: Within 5 minutes after delivery
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
mmol/L | -4.83 (2.47) | -8.23 (6.71)
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p = 0.201, Kruskal-Wallis

6. Other Pre Specified Outcome: Number of Participants With Intraoperative Hypotension
Time Frame: Intraoperatively from spinal placement till 10 minutes after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
Participants | 8 | 4
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p > 0.999, Fisher Exact

7. Other Pre Specified Outcome: Number of Participants With Intraoperative Nausea
Time Frame: Intraoperatively from time of spinal placement until end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
Participants | 5 | 3
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p = 0.962, Fisher Exact

8. Other Pre Specified Outcome: Number of Participants With Intraoperative Vomiting
Time Frame: Intraoperatively from time of spinal placement until end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 9 | 4
Participants | 2 | 1
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Other; p > 0.999, Fisher Exact

ADVERSE EVENTS:
Time Frame: From admission to discharge (no more than a few days).
Arm/Group | Phenylephrine | Ephedrine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 0/9 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes